CLINICAL TRIAL: NCT02269631
Title: Legume Diet Satiety and Weight Loss Pilot Study
Brief Title: Legume Diet Satiety Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Terry Hartman, Terry Hartman PhD, MPH, RD, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00075830
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Colorectal Carcinoma
Keywords: Weight loss; Epidemiology; Nutrition
MeSH Terms: conditions — Obesity; Colorectal Neoplasms; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Legume diet group (Experimental): Meals will include approximately 1 ½ cups of cooked legumes, such as pinto, baked and navy beans as part of your 2 daily main dishes (lunch and dinner) and additional foods and snacks, preferably from the recommended healthy foods list. The smartpill will be administered at the end of the study.
  Interventions: Behavioral: Legume diet group; Device: Smartpill; Other: legumes
- Control diet group (Active Comparator): Meals will be healthy, typical American foods (without legumes) for 2 daily main dishes and additional foods and snacks, preferably from the recommended healthy foods list.The smartpill will be administered at the end of the study.
  Interventions: Behavioral: Control diet group; Device: Smartpill

INTERVENTIONS:
Behavioral: Legume diet group — about 1 1/2 cups of legumes included in lunch and dinner meals
  Arms: Legume diet group
Behavioral: Control diet group — no legumes in lunch or dinner meals
  Arms: Control diet group
Device: Smartpill — to assess how long food takes to pass through the digestive system
Other: legumes — about 1 1/2 cups of legumes included in lunch and dinner meals
  Arms: Legume diet group

SUMMARY:
This pilot study is designed to test the effects of a high legume (dried bean) diet on hunger and other indicators of health over the course of eight weeks, compared to a more conventional healthy diet.

DETAILED DESCRIPTION:
The goal of the currently proposed study is to conduct a randomized controlled feeding pilot study within a more diverse population also at high risk for colorectal carcinoma (CRC) to evaluate whether a high-legume diet will result in increased satiety and in turn will facilitate reduced energy intake and weight loss compared to a control diet provided under similar conditions. In addition, explore potential beneficial effects of the high-legume diet on gastric emptying and circulating levels of appetite-regulating hormones and other biomarkers. Dietary behaviors that are even moderately more satiating over time have the potential to enhance weight loss and could lead to a significant public health impact among populations at high risk for colorectal carcinoma (CRC) and other chronic diseases.

Towards the end of the study, the participants will do an additional test, looking at how long food takes to pass through the digestive system using a SmartPill capsule. The SmartPill is a pill about the size of a large multivitamin that can measure pH, pressure, and temperature changes, which it uses to assess where in the digestive tract it is. The participant swallows the pill, and carries around a receiver that is about the size of a deck of cards for the next 3-5 days. The SmartPill is expelled, and the receiver notifies the participant that they can return the receiver to the study personnel.

ELIGIBILITY:
Inclusion Criteria:

* BMI overweight-obese: 25.0-40 kg/m2
* Colonoscopy within the last two years that found ≥1 adenoma
* English speaking
* Ambulatory, able to come to either food distribution site to pick up food and participate in clinical examinations and laboratory tests

Exclusion Criteria:

* Serious medical condition (e.g., cancer, heart disease, kidney disease, diabetes)
* History of CRC, bowel resection, polyposis syndrome, or inflammatory bowel disease
* Smoked regularly in the past year
* Dietary restrictions substantially limiting compliance or vegetarian or Vegan diet
* Planning on changing diet or exercise behavior in the next 6 months
* Regular use of medication that may alter inflammation markers, insulin, glucose, or gut function (i.e. regular use of non-steroidal anti-inflammatory medication, insulin therapy, steroid therapy, or antibiotics)

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry J Hartman, PhD, MPH, RD, Principal Investigator — Rollins School of Public Health, Emory University
Locations (2):
- United States (2):
  - Morehouse, Atlanta, Georgia
  - Emory ACTSI, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Legume Diet Group | Control Diet Group
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Legume Diet Group | Control Diet Group | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Evaluate the effects of a high-legume diet compared to a control diet with a similar macronutrient profile on weight change in a randomized controlled feeding study.
Time Frame: Baseline to 8 weeks
Measure: Median (Full Range); unit: lbs
Arm/Group | Legume Diet Group | Control Diet Group
Number analyzed (Participants) | 7 | 5
lbs | 9.2 [5.3 to 18.7] | 6.6 [6.2 to 11.4]

2. Secondary Outcome: Gastric Emptying Time
Description: Compare the effects of the high-legume and control diets on gastric emptying time
Time Frame: 8 weeks
Measure: Median (Full Range); unit: hours
Arm/Group | Legume Diet Group | Control Diet Group
Number analyzed (Participants) | 7 | 5
hours | 25.8 [20.8 to 56.8] | 53.8 [9.3 to 95.4]

3. Secondary Outcome: Change in Plasma Insulin Level (Biomarker of Appetite Regulation)
Description: Compare the effects of the high-legume and control diets on plasma insulin level in a meal response time (30 min) course experiment.
Time Frame: Baseline to 8 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Legume Diet Group | Control Diet Group
Number analyzed (Participants) | 7 | 5
mg/dl | -9.9 [-75 to 55] | 5.9 [-58 to 70]

4. Secondary Outcome: Energy Intake
Description: Compare the effects of the high-legume and control diets on self-reported dietary intake measured by telephone 24-hour dietary recalls.
Time Frame: Baseline to 8 weeks
Population: Data were collected but not analyzed due to a lack of funding.
Arm/Group | Legume Diet Group | Control Diet Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Satiety
Description: Use self-reported satiety questionnaire to compare short-term responses to test meals.
Time Frame: Time course response at baseline and 8 weeks
Population: Data were collected but not analyzed due to a lack of funding.
Arm/Group | Legume Diet Group | Control Diet Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Legume Diet Group | Control Diet Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02269631/Prot_SAP_000.pdf